CLINICAL TRIAL: NCT07176845
Title: Exploring Multidimensional Trajectories in People With Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); University of Zurich (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Stefan Schmid, Prof. Dr., Bern University of Applied Sciences
Other Study IDs: 2024-01927; 220434 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Low Back Pain; Chronic Low Back Pain (CLBP)
Keywords: low back pain; LBP; spinal motion; spine; disability; motor behavior; physical activity; pain-related fear; psychological factors
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute low back pain: Patients with an acute low back pain episode (<3 months of low back pain upon study enrollment)
  Interventions: Other: Observational
- Chronic low back pain: Patients with chronic low back pain (>3 months of low back pain upon study enrollment)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This study is observational of nature: multidimensional data is collected and no interventional is imposed

SUMMARY:
Low back pain (LBP) is a major health problem in Switzerland and worldwide. Globally, LBP remains the leading cause of years lived with disability and its incidence and associated socioeconomic consequences are predicted to increase in the coming decades. In Switzerland, the condition is one of the most commonly reported physical complaints and negatively affects quality of life, resulting in significant personal burden and personal financial burden. LBP also generates enormous socioeconomic costs, with both direct and indirect costs estimated to reach billions of Swiss francs in Switzerland annually. Therefore, it is essential that LBP prevention, diagnosis, and management are improved.

LBP is a multifactorial condition. Social, psychological and biophysical factors, along with comorbidities and genetic factors, influence LBP development and associated disability. In individuals with LBP, psychological factors, such as pain catastrophizing, are associated with higher pain intensity and developing chronic LBP and the associated disability. Among biophysical factors, altered spinal motor behaviour (e.g. smaller trunk movement amplitude) and reduced physical activity have been observed in LBP patients and suggested to influence LBP. However, exactly how all these factors influence LBP and how they are interrelated remains unclear. In particular, the effect of altered spinal motor behaviour on LBP is not understood. However, altered motor behaviour could play an important role in changing LBP and related disability. Therefore, improving our understanding of the patterns of spinal motor behaviour and the interrelationships with other factors in LBP would increase our understanding of LBP progression and could help improve LBP management.

This study consists of a 6-month prospective longitudinal cohort observation of spinal motor behavior, physical activity, psychological factors, pain intensity, and disability in LBP patients (300 acute, 300 chronic LBP). Data collection will occur remotely and the frequency of repeated measures will be daily or weekly, depending on the measure. A custom smart-phone application will be used by participants to collect data on spinal motor behavior, psychological factors, pain intensity, and disability. Physical activity will be monitored using a wearable physical activity tracker.

Established trajectories of motor behavior will be investigated for potential interrelations with trajectories of other parameters (e.g. pain, psychological factors, and disability), to explore potential causal effects. In addition, risk factors or predictive factors for certain trajectories of motor behavior and other parameters will be identified. As such, this study will allow us to investigate the temporality of these relationships and identify LBP, and in particular spinal motor behavior, phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* have low back pain (rate their LBP with an intensity of >0 on a 0-10 numerical pain rating scale at enrollment)
* 18 years old or older
* be proficient in German, French, or English
* own a smartphone that is able to run either Android or iOS (iPhone) apps
* own a smartphone that includes accelerometer and gyroscope sensors

Exclusion Criteria:

* diagnosis of a specific LBP etiology (e.g. fracture, tumoral process, radiculopathy with evidence of neurological deficit or cauda equina)
* history of previous spinal fusion surgery, which would influence on motor behavior
* presence of any other medical conditions (pathologies, diseases, comorbidities, injuries, surgeries or painful conditions) that could jeopardize the patients' safety, prevent them from performing the spinal motion measurements safely (e.g., risk of falls due to frailty), or influence spinal motion (e.g., Parkinson's disease, stroke)
* inability to follow procedures
* inability to give consent (e.g. dementia)
* owner of a smartphone, not able to run an Android or iPhone application
* owner of a smartphone without accelerometer and gyroscope sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from ambulatory medical, physiotherapy and rehabilitation clinics in northern, central and western Switzerland (cantons: Bern, Zürich, Basel, Aargau, Luzern, Zug, Schwyz, Vaud, Fribourg, Wallis, and Neuchâtel).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Spinal motion: maximum movement amplitude | Up to 25 weeks from enrollment.
  Spine motion is recorded during multiple repetitions of several clinically relevant motions (trunk flexion, trunk extension, left/right trunk lateral flexion while standing), as well as a functional motion (picking up a lightweight object from the floor). The motion is measured using the internal inertial sensors of the patient's smartphone.
  The first main variable of interest is maximum movement amplitude (unit: degrees).
  Frequency of measurement: weekly during the 25-week study period.
Spinal motion: maximum/average movement velocity | Up to 25 weeks from enrollment.
  Spine motion is recorded during multiple repetitions of several clinically relevant motions (trunk flexion, trunk extension, left/right trunk lateral flexion while standing), as well as a functional motion (picking up a lightweight object from the floor). The motion is measured using the internal inertial sensors of the patient's smartphone.
  The second main variable of interest is maximum/average movement velocity (unit: degrees/second).
  Frequency of measurement: weekly during the 25-week study period.
Movement-evoked low back pain | Up to 25 weeks from enrollment.
  Movement-evoked low back pain (pain during movement) will be scored by patients on an 11-point numerical pain rating scale (0-10; whole-point, with 0 being 'no pain' and 10 'the worst pain you can imagine'), for each spinal motion separately, directly after performing each movement.
  Frequency of measurement: weekly during the 25-week study period.
Psychological factors: movement pain-related fear | Up to 25 weeks from enrollment.
  Pain-related fear will be assessed for each movement being measured, using an 11-point numerical rating scale (0-10; whole-point), with 0 being 'not harmful at all' and 10 'extremely harmful' (adapted from Photograph Series of Daily Activities-Short Electronic Version; PHODA-SeV).
  Frequency of measurement: weekly during the 25-week study period.
Psychological factors: task-specific pain-related fear | Up to 25 weeks from enrollment.
  Item four from the Photograph Series of Daily Activities-Short Electronic Version (PHODA-SeV), which shows a person lifting a pot, will be used to assess task-specific pain-related fear. Participants rate their fear on an 11-point numerical rating scale (0-10; whole-point), with 0 being 'not harmful at all' and 10 'extremely harmful'.
  Frequency of measurement: weekly during the 25-week study period.
Psychological factors: fear avoidance beliefs related to physical activity | Up to 25 weeks from enrollment.
  The physical activity subscale of the Fear-Avoidance Beliefs Questionnaire (FABQ) will be used to assess fear avoidance beliefs related to physical activity. Frequency of measurement: weekly during the 25-week study period.
Psychological factors: pain catastrophizing | Up to 25 weeks from enrollment.
  Pain catastrophizing will be assessed using the Daily Pain Catastrophizing Scale (Daily PCS). Frequency of measurement: weekly during the 25-week study period.
Psychological factors: self-efficacy | Up to 25 weeks from enrollment.
  Self-efficacy will be measured using the 2-item short form of the Pain Self-Efficacy Questionnaire (PSEQ-2). Frequency of measurement: weekly during the 25-week study period.
Psychological factors: stress | Up to 25 weeks from enrollment.
  Stress across the last 24 hours will be assessed using the 11-point stress numerical rating scale (0-10, whole-point, with 0 being 'no stress' and 10 being 'worst stress imaginable'). Frequency of measurement: weekly during the 25-week study period.
Physical activity: heart rate | Up to 25 weeks from enrollment.
  Physical activity is measured continuously using a well-established, wrist-worn activity tracker.
  The first main variable of interest is heart rate (unit: beats per minute). Frequency of measurement: continuously during the 25-week study period.
Physical acitivity: step count | Up to 25 weeks from enrollment.
  Physical activity is measured continuously using a well-established, wrist-worn activity tracker.
  The second main variable of interest is step count (unit: number of steps). Frequency of measurement: continuously during the 25-week study period.
Low back pain intensity | Up to 25 weeks from enrollment.
  Average low back pain intensity, in the last 24 hours, will be scored by patients on an 11-point numerical pain rating scale (0-10; whole-point), with 0 being 'no pain' and 10 'the worst pain you can imagine'.
  Frequency of measurement: daily during the 25-week study period.
Disability: general level of disability (1) | Up to 25 weeks from enrollment.
  General level of disability will be rated by patients using an 11-point numerical rating scale (0-10; whole-point, with 0 'not at all', 5 'moderate limitation', 10 'totally limited').
  Frequency of measurement: weekly during the 25-week study period.
Disability: general level of disability (2) | Up to 25 weeks from enrollment.
  General level of disability will also be rated by patients using the Roland-Morris Disability Questionnaire (RMDQ).
  Frequency of measurement: 6-weekly during the 25-week study period.
Disability: lift-specific disability | Up to 25 weeks from enrollment.
  The LBP impact on the patient's ability to lift over the past 24 hours will be assessed using one single-item question and rated using an 11-point numeric rating scale (0-10; whole-point, with 0 being 'not al all', 5 'moderate limitation', 10 'totally limited'). Frequency of measurement: weekly during the 25-week study period.

SECONDARY OUTCOMES:
Patient demographics: sex | At enrollment
  Data on sex (female, male, intersex) will be collected using a questionnaire.
Patient demographics: gender | At enrollment
  Data on gender (woman, man, non-binary, a term not listed, I am questioning/not sure) will be collected using a questionnaire.
Patient demographics: occupational status | At enrollment
  Data on occupational status will be collected using a questionnaire.
Patient demographics: occupation | At enrollment
  Data on current or recent occupation will be collected using a questionnaire.
Patient demographics: work satisfaction | At enrollment
  Data on work satisfaction (very unsatisfied; unsatisfied; neutral; satisfied; very satisfied; this is not relevant to me) will be collected using a questionnaire.
Patient demographics: work expectation | At enrollment
  Data on work expectation ('I think I will be able to do my regular job, without any restrictions, 4 weeks from now' and 'I think I will be able to do my regular job, without any restrictions, 3 months from now'; on a 7-point scale, 0-6 with 0 being 'unlikely' and 6 'definitely') will be collected using a questionnaire.
Patient demographics: highest education | At enrollment
  Data on highest education will be collected using a questionnaire.
Patient anthropometry: body mass | At enrollment
  Patient body mass (unit: kg) will be collected using a questionnaire
Patient anthropometry: height | At enrollment
  Patient height (unit: m) data will be collected using a questionnaire
Basic low back pain history: duration | At enrollment
  Data on duration of low back pain symptoms will be collected using a questionnaire
Basic low back pain history: other | At enrollment
  Data on location and previous episodes of low back pain symptoms, and other diagnoses or previous surgeries will be collected using a questionnaire.
Low back pain beliefs | At enrollment
  Data on low back pain beliefs will be collected using the BackPAQ questionnaire.
Basic medical status: smoking status | At enrollment
  Data on smoking status (yes; no, not anymore; no, never) will be collected using a questionnaire
Basic medical status: comorbidities | At enrollment
  Data on comorbidities will be collected using a questionnaire
Basic medical status: anxiety | At enrollment
  Data on anxiety will be collected using a questionnaire on an 11-point scale (0-10, whole-point) numerical rating scale, with 0 being 'not at all' and 10 'quite anxious'.
Basic medical status: depression | At enrollment
  Data on depression will be collected using a questionnaire on an 11-scale (0-10, whole-point) numerical rating scale, with 0 being 'never' and 10 'all the time'.
Basic medical status: stress | At enrollment
  Data on stress will be collected using the perceived stress scale 4 questionnaire, with for each of the four questions a 5-point scale (0-4, whole-point, with 0 being 'never' and 4 'very often').
Basic medical status: medication and treatment | At enrollment
  Data on medication as well as previous and current treatment will be collected using a questionnaire
Basic medical status: neuropathic pain | At enrollment
  Data on neuropathic pain symptoms will be collected using the first two questions of neuropathic pain diagnosis questionnaire (DN4). For both questions, participants select symptoms from a list, with each selected symptom scored as +1, with a total score of larger than or equal to 3 indicating neuropathic pain.

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored in a private repository during the project and, upon its completion, will be made publicly available on the Swiss-based data management portal OLOS under a CC0 license. OLOS was chosen because it supports the FAIR principles and offers robust long-term preservation features. Data not publicly released on OLOS will be accessible upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol, including the statistical analysis plan, will be published in a scientific journal before the end of the data collection. All other publicly made data will be available indefinitely upon completion of the project.
Access Criteria: Everyone via OLOS or upon reasonable request.

REFERENCES:
- [Background] Christe G, Benaim C, Jolles BM, Favre J. Changes in spinal motor behaviour are associated with reduction in disability in chronic low back pain: A longitudinal cohort study with 1-year follow-up. Eur J Pain. 2024 Aug;28(7):1116-1126. doi: 10.1002/ejp.2245. Epub 2024 Feb 1. PMID 38299715
- [Background] Moissenet F, Armand S, Genevay S. Measurement properties of 72 movement biomarkers aiming to discriminate non-specific chronic low back pain patients from an asymptomatic population. Sci Rep. 2023 Apr 20;13(1):6483. doi: 10.1038/s41598-023-33504-5. PMID 37081110
- [Background] Kongsted A, Kent P, Axen I, Downie AS, Dunn KM. What have we learned from ten years of trajectory research in low back pain? BMC Musculoskelet Disord. 2016 May 21;17:220. doi: 10.1186/s12891-016-1071-2. PMID 27209166
- [Background] Martinez-Calderon J, Jensen MP, Morales-Asencio JM, Luque-Suarez A. Pain Catastrophizing and Function In Individuals With Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis. Clin J Pain. 2019 Mar;35(3):279-293. doi: 10.1097/AJP.0000000000000676. PMID 30664551
- [Background] Moissenet F, Rose-Dulcina K, Armand S, Genevay S. A systematic review of movement and muscular activity biomarkers to discriminate non-specific chronic low back pain patients from an asymptomatic population. Sci Rep. 2021 Mar 12;11(1):5850. doi: 10.1038/s41598-021-84034-x. PMID 33712658
- [Background] Buchbinder R, Underwood M, Hartvigsen J, Maher CG. The Lancet Series call to action to reduce low value care for low back pain: an update. Pain. 2020 Sep;161 Suppl 1(1):S57-S64. doi: 10.1097/j.pain.0000000000001869. No abstract available. PMID 33090740
- [Background] Wieser, S., Tomonaga, Y., Riguzzi, M., Fischer, B., Telser, H., Pletscher, M., Eichler, K., Trost, M., & Schwenkglenks, M. (2014). Die Kosten der nichtübertragbaren Krankheiten in der Schweiz: Schlussbericht. Zürich Open Repository and Archive. https://doi.org/10.5167/UZH-103453
- [Background] Rheumaliga Schweiz. (2020). Rückenreport Schweiz 2020. https://www.rheumaliga.ch/blog/2020/rueckenreport-2020
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Bundesamt für Statistik. (2023). Schweizerische Gesundheitsbefragung 2022. Übersicht (No. BFS-Nummer 213-2201; S. 1-28). Bundesamt für Statistik. https://www.bfs.admin.ch/asset/de/28465284
- [Background] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833
- See also: Swiss National Science Foundation - Project page — https://data.snf.ch/grants/grant/220434